CLINICAL TRIAL: NCT06902558
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of ABBV-CLS-628 in Adult Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: A Study to Assess Adverse Events and Effectiveness of IntraVenous Infusions of ABBV-CLS-628 in Adult Participants With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Acronym: ANCHOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M25-147; 2024-517143-31-00 (Other: EU CT)
Record Dates: First submitted 2025-03-25; First posted 2025-03-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal Dominant Polycystic Kidney Disease (ADPKD); ABBV-CLS-628
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ABBV-CLS-628 Dose A (Experimental): Participants will receive ABBV-CLS-628 Dose A every 4 weeks for 92 weeks.
  Interventions: Drug: ABBV-CLS-628
- ABBV-CLS-628 Dose B (Experimental): Participants will receive ABBV-CLS-628 Dose B every 4 weeks for 92 weeks.
  Interventions: Drug: ABBV-CLS-628
- ABBV-CLS-628 Dose C (Experimental): Participants will receive ABBV-CLS-628 Dose C every 4 weeks for 92 weeks.
  Interventions: Drug: ABBV-CLS-628
- Placebo (Placebo Comparator): Participants will receive ABBV-CLS-628 Placebo every 4 weeks for 92 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABBV-CLS-628 — IntraVenous Infusion
  Arms: ABBV-CLS-628 Dose A; ABBV-CLS-628 Dose B; ABBV-CLS-628 Dose C
Drug: Placebo — IntraVenous Infusion
  Arms: Placebo

SUMMARY:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the most common genetic cause of kidney disease that causes fluid-filled cysts to develop in the kidneys. The purpose of this study is to assess the safety and efficacy of ABBV-CLS-628 for the treatment of ADPKD in adult participants.

ABBV-CLS-628 is an investigational drug being developed for the treatment of ADPKD. Participants are placed in 1 of 4 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 4 chance that participants will be assigned to placebo. Around 240 adult participants with ADPKD will be enrolled at approximately 100 sites worldwide.

Participants will receive IntraVenous ABBV-CLS-628 or placebo every 4 weeks for 92 weeks. Participants will be followed for up to 15 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care . Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Autosomal Dominant Polycystic Kidney Disease (ADPKD) Class 1C, 1D, or 1E based on the Mayo Clinic Imaging Classification of ADPKD.
* Estimated glomerular filtration rate (eGFR) >= 30 mL/min/1.73 m^2 and < 90 mL/min/1.73 m^2, using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at Screening.

Exclusion Criteria:

* Current interventions to treat ADPKD such as non-approved medications or lifestyle modifications.
* Any exclusionary medical diseases, disorders, or conditions as described in the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative Rate of Change from Baseline in Total Kidney Volume (TKV) | Week 96
  TKV will be determined from manual contours of the kidneys on 3D magnetic resonance imaging (MRI), performed by imaging specialists and verified by independent radiologists with expertise in Autosomal Dominant Polycystic Kidney Disease (ADPKD).
Number of Participants with Adverse Events (AEs) | Up to approximately 118 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Absolute Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline | Week 96
  eGFR will be measured using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine equation (2021) and CKD-EPI Creatinine-Cystatin equation (2021).
Cumulative Rate of Change from Baseline in Total Kidney Volume (TKV) | Week 48
  TKV will be determined from manual contours of the kidneys on 3D magnetic resonance imaging (MRI), performed by imaging specialists and verified by independent radiologists with expertise in Autosomal Dominant Polycystic Kidney Disease (ADPKD).
Absolute Change in eGFR From Baseline | Week 48
  eGFR will be measured using the CKD-EPI Creatinine equation (2021) and CKD-EPI Creatinine-Cystatin equation (2021).
Time From Randomization to the First Occurrence of Clinical Progression to End-Stage Kidney Disease (ESKD) or >= 40% Decline in eGFR | Up to Week 96
  Defined as initiation of renal replacement therapy (RRT) or kidney transplantation, or a confirmed decline in eGFR of 40% or more from baseline, sustained for at least 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (75):
- United States (35):
  - National Institute of Clinical Research - Garden Grove /ID# 271418, Garden Grove, California
  - Valiance Clinical Research - Huntington Park /ID# 270634, Huntington Park, California
  - Academic Medical Research Institute - Los Angeles /ID# 270502, Los Angeles, California
  - UC Irvine Medical Center /ID# 270811, Orange, California
  - University Of California, San Francisco /ID# 270326, San Francisco, California
  - Yale University School of Medicine /ID# 270675, New Haven, Connecticut
  - Horizon Research Group - Coral Gables /ID# 270857, Coral Gables, Florida
  - South Florida Research Institute /ID# 270848, Fort Lauderdale, Florida
  - Nature Coast Clinical Research - Inverness /ID# 270875, Inverness, Florida
  - Mayo Clinic Hospital Jacksonville /ID# 271011, Jacksonville, Florida
  - Panax Clinical Research /ID# 270851, Miami, Florida
  - Infigo Clinical Research /ID# 270844, Sanford, Florida
  - Emory University School Of Medicine - Atlanta /ID# 271947, Atlanta, Georgia
  - CARE-Boise Kidney /ID# 270628, Boise, Idaho
  - CARE Institute - Idaho Falls /ID# 272005, Idaho Falls, Idaho
  - Northwestern University Feinberg School of Medicine /ID# 271409, Chicago, Illinois
  - University of Iowa /ID# 270492, Iowa City, Iowa
  - University of Kansas Medical Center /ID# 271946, Kansas City, Kansas
  - Tufts Medical Center /ID# 270323, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 271408, Boston, Massachusetts
  - University Of Michigan /ID# 270436, Ann Arbor, Michigan
  - St. Clair Nephrology /ID# 271445, Shelby, Michigan
  - Mayo Clinic Hospital Rochester /ID# 270428, Rochester, Minnesota
  - Washington University /ID# 271436, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai /ID# 271440, New York, New York
  - University of North Carolina at Chapel Hill /ID# 274800, Chapel Hill, North Carolina
  - Brookview Hills Research Associates /ID# 271449, Winston-Salem, North Carolina
  - Northeast Clinical Research Center /ID# 270838, Bethlehem, Pennsylvania
  - University of Pennsylvania /ID# 270301, Philadelphia, Pennsylvania
  - Nephrology Associates - Chattanooga - East Third Street /ID# 270701, Chattanooga, Tennessee
  - Knoxville Kidney Center /ID# 270706, Knoxville, Tennessee
  - Arlington Nephrology /ID# 270494, Arlington, Texas
  - Renal Disease Research Institute /ID# 270339, Fort Worth, Texas
  - University of Virginia /ID# 270329, Charlottesville, Virginia
  - Swedish Medical Center - Seattle /ID# 270344, Seattle, Washington
- Australia (4):
  - Westmead Hospital /ID# 271156, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 271224, Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 273114, Adelaide, South Australia
  - Fiona Stanley Hospital /ID# 271173, Murdoch, Western Australia
- Belgium (3):
  - Cliniques Universitaires UCL Saint-Luc /ID# 270635, Brussels, Brussels Capital
  - UZ Leuven /ID# 270638, Leuven, Vlaams-Brabant
  - CHU de Liege /ID# 270631, Liège
- France (5):
  - Hopital Edouard Herriot /ID# 271142, Lyon, Auvergne-Rhône-Alpes
  - CHU Brest - Hôpital de la Cavale Blanche /ID# 271114, Brest, Brittany Region
  - CHU Toulouse - Hôpital Rangueil /ID# 271138, Toulouse, Occitanie
  - Hopital de la Conception /ID# 271152, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hopital Universitaire Necker Enfants Malades /ID# 271146, Paris, Île-de-France Region
- Germany (4):
  - TUM Klinikum rechts der Isar /ID# 271522, Munich, Bavaria
  - Medizinische Hochschule Hannover /ID# 270938, Hanover, Lower Saxony
  - Universitaetsklinikum Koeln /ID# 270937, Cologne, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 270935, Berlin
- Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 271563, Rome, Roma, Italy
- Japan (4):
  - Hokkaido University Hospital /ID# 271385, Sapporo, Hokkaido
  - National Hospital Organization Kyoto Medical Center /ID# 271782, Kyoto, Kyoto
  - Juntendo University Hospital /ID# 271722, Bunkyo-ku, Tokyo
  - National Hospital Org Chiba Medical Center Chibahigashi National Hospital /ID# 272022, Chiba
- Netherlands (3):
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk /ID# 271247, Dordrecht, South Holland
  - Lumc /Id# 271844, Leiden, South Holland
  - Universitair Medisch Centrum Groningen /ID# 271249, Groningen
- Portugal (5):
  - Unidade Local de Saude de Almada-Seixal, EPE /ID# 271257, Almada, Setúbal District
  - 2CA-Braga, Hospital de Braga /ID# 271258, Braga
  - Unidade Local de Saude do Algarve, EPE /ID# 271819, Faro
  - Unidade Local de Saude de Sao Jose, EPE /ID# 271255, Lisbon
  - Unidade Local de Saude de Lisboa Ocidental, EPE /ID# 271261, Lisbon
- South Korea (5):
  - Pusan National University Hospital /ID# 271429, Busan, Busan Gwang Yeogsi
  - Keimyung University Dongsan Hospital /ID# 272455, Daegu, Gyeongsangbuk-do
  - Seoul National University Hospital /ID# 271331, Seoul, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 271227, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 271329, Seoul, Seoul Teugbyeolsi
- Spain (6):
  - Hospital Universitari de Bellvitge /ID# 270489, L'Hospitalet de Llobregat, Barcelona
  - Fundacio Puigvert /ID# 270491, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 270918, Granada
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 270485, Madrid
  - Hospital Universitario 12 de Octubre /ID# 270829, Madrid
  - Hospital Clínico Universitario de Valencia /ID# 270837, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Cortinovis M, Perico N, Remuzzi G. The Need for Novel Therapeutic Directions in Autosomal Dominant Polycystic Kidney Disease Patient Care. Clin J Am Soc Nephrol. 2025 Dec 5. doi: 10.2215/CJN.0000000975. Online ahead of print. PMID 41348481
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-147